CLINICAL TRIAL: NCT03965442
Title: Effects of Intraoperative Esmolol on Post-mastectomy Pain Syndrome: a Cross-sectional Study
Brief Title: Effects of Intraoperative Esmolol on Post-mastectomy Pain Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, Preceptor correspondent for anesthesiology residency, Hospital de Base
Other Study IDs: Post-mastectomy pain
Record Dates: First submitted 2019-02-21; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Post-mastectomy Pain Syndrome
Keywords: Post-mastectomy Pain Syndrome; Esmolol; Perioperative
MeSH Terms: interventions — esmolol

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Patients who underwent mastectomy under standard general anesthesia
  Patients in placebo group received general balanced inhaled anesthesia with sevoflurane and remifentanil and a saline 0,9% infusion pump.
  Interventions: Drug: Control
- Esmolol: Patients in esmolol group received general balanced inhaled anesthesia with sevoflurane and a bolus infection of esmolol 500 mgc/kg followed by a continuous infusion of esmolol 100 mcg/kg/min
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Control — Patients who underwent mastectomy under standard general anesthesia
  Groups: Control
Drug: Esmolol — Patients who underwent mastectomy under general anesthesia with esmolol infusion
  Groups: Esmolol

SUMMARY:
Chronic postoperative pain is an entity that is usually neglected by anesthetists, but several studies show that the choice of anesthetic technique may interfere with this prevalence. Esmolol is a selective beta-blocker of ultra fast duration that has been studied as a perioperative venous adjuvant with antihyperalgesic and opioid sparing action. The investigators ventured the possibility of this anti-hyperalgesic effect attenuating the chronic pain syndrome post-mastectomy.

ELIGIBILITY:
Inclusion Criteria:

- Patients previously submitted to the study Analgesic Effect of Intraoperative Esmolol in Mastectomies: a randomized placebo controlled trial

Exclusion Criteria:

* Patient aged less than 18 years and over 65 years;
* Patients who refuse to participate in the study;
* Patients with pulmonary disease;
* Patients with cardiac, renal or hepatic disease;
* Use of psychoactive drug;
* Patients with sinus bradycardia;
* Pregnant women;
* Patients with allergy to dipyrone, morphine;
* Patients with chronic pain prior to the surgical procedure;
* Patients with neurological disorders;
* Patients undergoing surgical resurfacing

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously submitted to the study Analgesic Effect of Intraoperative Esmolol in Mastectomies: a randomized placebo controlled trial, will be submitted to a questionnaire of adapted from DNS4.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-mastectomy chronic pain syndrome | Through study completion, an average of 6 to 9 month
  Incidence analysis using a questionnaire applied to patients in the late postoperative period.

SECONDARY OUTCOMES:
Assess the intensity of pain: Pain Scores on the Visual Analog Scale | Through study completion, an average of 6 to 9 month
  Pain Scores on the Visual Analog Scale, from zero to 10: 0 being represented by absence of pain and 10 being the worst possible pain
Identify possible risk factors | Through study completion, an average of 6 to 9 month
  Incidence analysis using a questionnaire applied to patients in the late postoperative period.
Stratify the possible types of pain | Through study completion, an average of 6 to 9 month
  Application of a questionnaire to identify the characteristics of pain (Neuropatic or non-neuropatic pain)

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonça, MD, Principal Investigator — Hospital de Base do Distrito Federal
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919